CLINICAL TRIAL: NCT04201873
Title: Phase I Surgical Trial to Evaluate Early Immunologic Pharmacodynamic Parameters for the PD-1 Antibody Pembrolizumab With Autologous Tumor Lysate-Pulsed Dendritic Cell Vaccination in Patients With Surgically Accessible Recurrent/Progressive Glioblastoma
Brief Title: Pembrolizumab and a Vaccine (ATL-DC) for the Treatment of Surgically Accessible Recurrent Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Merck Sharp & Dohme LLC (Industry); Phase One Foundation (Other); Oncovir, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-001090; NCI-2019-07994 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-001090 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — pembrolizumab; poly ICLC

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (pembrolizumab, ATL-DC, poly ICLC) (Experimental): Beginning 14 days prior to scheduled surgery, patients receive pembrolizumab IV over 30 minutes. After surgery, patients receive pembrolizumab IV over 30 minutes on day 1. Cycle repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive ATL-DC ID with poly ICLC IM every 2 weeks for up to 3 doses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Dendritic Cell Tumor Cell Lysate Vaccine; Biological: Pembrolizumab; Drug: Poly ICLC
- Group B (placebo, ATL-DC, poly ICLC) (Active Comparator): Beginning 14 days prior to scheduled surgery, patients receive placebo IV. After surgery, patients receive placebo IV on day 1. Cycle repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive ATL-DC ID with poly ICLC IM every 2 weeks for up to 3 doses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Dendritic Cell Tumor Cell Lysate Vaccine; Other: Placebo Administration; Drug: Poly ICLC

INTERVENTIONS:
Biological: Dendritic Cell Tumor Cell Lysate Vaccine — Given ID
  Other Names: DC tumor cell lysate vaccine; dendritic cell-pulsed tumor cell lysate vaccine
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
  Arms: Group A (pembrolizumab, ATL-DC, poly ICLC)
Other: Placebo Administration — Given IV
  Arms: Group B (placebo, ATL-DC, poly ICLC)
Drug: Poly ICLC — Given IM
  Other Names: Hiltonol; Poly I:Poly C with Poly-L-Lysine Stabilizer; poly-ICLC; PolyI:PolyC with Poly-L-Lysine Stabilizer; Polyinosinic-Polycytidylic Acid Stabilized with Polylysine and Carboxymethylcellulose; Polyriboinosinic-Polyribocytidylic Acid-Polylysine Carboxymethylcellulose; Stabilized Polyriboinosinic/Polyribocytidylic Acid

SUMMARY:
This phase I trial studies the side effects and how well of pembrolizumab and a vaccine therapy (ATL-DC vaccine) work in treating patients with glioblastoma that has come back (recurrent) and can be removed by surgery (surgically accessible). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Vaccines, such as ATL-DC vaccine, may help the body build an effective immune response to kill tumor cells. Giving pembrolizumab and ATL-DC vaccine may work better in treating patients with glioblastoma compared to ATL-DC alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the influence of pembrolizumab on the cell cycle-related genetic signature within the tumor microenvironment of progressive/recurrent glioblastoma.

II. To evaluate the influence of adjuvant autologous tumor lysatepulsed dendritic cell (ATL-DC) vaccination on peripheral T cell responses.

III. To evaluate the safety and tolerability of pembrolizumab and ATL-DC vaccination in progressive/recurrent glioblastoma.

SECONDARY OBJECTIVES:

I. To estimate the 6 month progression-free survival (PFS6) based on Response Assessment in Neuro-Oncology (RANO) criteria in patients treated on both arms of the clinical trial.

II. To calculate the overall survival of recurrent glioblastoma patients treated on both arms of the clinical trial.

EXPLORATORY OBJECTIVES:

I. To evaluate the associations between exploratory biomarkers, clinical outcomes, and adverse events which include:

Ia. Estimating the correlation of quantitative assessments of tumor infiltrating lymphocyte (TIL) density or the interferon (IFN) gamma-associated genetic signature with clinical responses to pembrolizumab and ATL-DC in recurrent glioblastoma patients.

Ib. Estimating the efficacy of pembrolizumab and ATL-DC through PFS6, PFS and overall survival (OS) as defined by RANO.

Ic. Estimating the efficacy of pembrolizumab and ATL-DC through PFS6, PFS, and OS as defined by immunotherapy RANO (iRANO).

Id. Exploring whether oligoclonal T cell populations within tumor tissue are similarly expanded in peripheral blood after ATL-DC vaccination and/or pembrolizumab, and correlating with clinical responses.

Ie. Exploring whether changes in specific magnetic resonance imaging (MRI) parameters correlate with tumor and peripheral blood immune responses.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP A: Beginning 14 days prior to scheduled surgery, patients receive pembrolizumab intravenously (IV) over 30 minutes. After surgery, patients receive pembrolizumab IV over 30 minutes on day 1. Cycle repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive ATL-DC intradermally (ID) with poly ICLC intramuscularly (IM) every 2 weeks for up to 3 doses in the absence of disease progression or unacceptable toxicity.

GROUP B: Beginning 14 days prior to scheduled surgery, patients receive placebo IV. After surgery, patients receive placebo IV on day 1. Cycle repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive ATL-DC ID with poly ICLC IM every 2 weeks for up to 3 doses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically confirmed diagnosis of surgically accessible recurrent/progressive glioblastoma will be enrolled in this study
* Be at first or second relapse (Note: relapse is defined as progression following initial therapy, i.e., radiation +/- chemotherapy. For participants who had prior therapy for a low-grade glioma, the surgical diagnosis of a high-grade glioma will be considered the first relapse)
* Must be undergoing surgery that is clinically indicated, and eligible for resection with the expectation that the surgeon is able to resect at least 2 gram of tumor for lysate and research with low risk of inducing neurological injury
* A male participant must agree to use a contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period
* A female participant who has childbearing potential must have negative urine or serum pregnancy test 72 hrs prior to the first dose and be willing to use adequate method of contraception for course of study and 120 days after last dose
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial
* Have unequivocal evidence for contrast enhancing tumor progression by RANO criteria based on MRI scan within 14 days prior to randomization
* Have a minimum tumor size of 2 x 2 cm^2 based on MRI scan prior to surgery
* An interval of the following durations prior to randomization:

  * At least 28 days from prior surgical resection
  * At least 7 days from prior stereotactic biopsy
  * At least 12 weeks from prior radiotherapy, unless there is unequivocal histologic confirmation of tumor progression
  * At least 23 days from prior chemotherapy
  * At least 42 days from nitrosureas
* Have sufficient archival tumor tissue confirming glioblastoma or variants for submission following registration. The following amount of tissue is required: 1 formalin-fixed, paraffin embedded (FFPE) tissue block (preferred) or 10 FFPE ,unstained slides (5um thick)
* Have a Karnofsky performance status (KPS) >= 70
* Absolute neutrophil count (ANC) >= 1500/uL (uL=microliter) (collected within 14 days prior to the start of study treatment)
* Platelets >= 100 000/uL (collected within 14 days prior to the start of study treatment)
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L (collected within 14 days prior to the start of study treatment)

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance >= 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN (collected within 14 days prior to the start of study treatment) (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl])

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN (collected within 14 days prior to the start of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT[) =< 2.5 x ULN (=< 5 x ULN for participants with liver metastases) (collected within 14 days prior to the start of study treatment)
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants (collected within 14 days prior to the start of study treatment)
* aPTT =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (collected within 14 days prior to the start of study treatment)

Exclusion Criteria:

* A woman of childbearing potential (WOCBP) who has a positive urine pregnancy test within 72 hours prior to randomization. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137)
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to randomization

  * Note: Participants must have recovered from all adverse events (AEs) due to previous therapies to =< grade 1 or baseline. Participants with =< grade 2 neuropathy may be eligible
  * Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-central nervous system (CNS) disease
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus calmette-guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist) are live attenuated vaccines and are not allowed
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment

  * Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years

  * Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* Has known tumor primarily localized to the brainstem or spinal cord
* Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV)
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as hepatitis C virus [HCV] ribonucleic acid [RNA] is detected) infection. Note: no testing for hepatitis B and hepatitis C is required unless mandated by local health authority
* Has a known history of active TB (Bacillus tuberculosis)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Cell cycle-related signature | Up to 6 years
Expansion of T cell receptor (TCR) clones | Up to 6 years
  Two-sample T-test with Bonferroni adjustment will be used to compare the increase number of expanded TCR clones after dendritic cell (DC) vaccination with PD-1 blockade in Group A versus (vs) DC vaccination with a placebo in Group B.
Incidence of adverse events (AEs) | Up to 30 days post treatment
  Adverse events will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. All patients who receive any amount of pembrolizumab/placebo or ATL-DC vaccination will be evaluable for toxicity, serious adverse events (SAEs), and events of clinical interest (ECIs).

SECONDARY OUTCOMES:
6 month progression-free survival (PFS6) | At 6 months
  Efficacy will be measured by percent PFS6 as defined by Response Assessment in Neuro-Oncology (RANO) criteria. Kaplan-Meier (KM) curves and median estimates from the KM curves will be provided as appropriate. Percent PFS6 will be estimated from the KM curves and compared to historical controls.
Overall survival (OS) | Up to 6 years
  OS will be compared using log rank test.

OTHER OUTCOMES:
Biomarker analysis | Up to 6 years
  The association between biomarkers and clinical outcomes (PFS and OS) will be evaluated using Cox regression. Changes in markers pre- and post- treatment will be assessed using paired t-tests.
TIL (tumor infiltrating lymphocyte) density and TCR (T cell receptor) Clonality in the tumor quantitatively measured by next generation TCR sequencing | from baseline to surgery
  The differences of TIL density and TCR Clonality between the archival tumor (pre-treatment) and protocol tumor (post-neoadjuvant treatment) will be assessed using paired T-test, and the association between the changes in TIL density and TCR Clonality and clinical outcome (PFS and OS) will be evaluated using Cox regression.
TIL density and TCR Clonality in the peripheral blood quantitatively measured by next generation TCR sequencing | from baseline to surgery and post surgery treatment period, up to 24 months
  The changes of TIL density and TCR Clonality in the peripheral blood from samples collected prior to neoadjuvant treatment and samples collected post-neoadjuvant treatment at each MRI visit will be assessed using paired T-test, and the association between the changes in TIL density and TCR Clonality and clinical outcome (PFS and OS) will be evaluated using Cox regression.
gene expression signature and somatic mutations in the tumor measured by RNA Seq and nano string IO360 | from baseline to surgery
  The differences of gene expression signature and somatic mutations between the archival tumor (collected pre-treatment) and protocol tumor (collected post-neoadjuvant treatment) will be assessed using paired T-test, and the association between the changes in the cell cycle related gene expression signature and clinical outcome (PFS and OS) will be evaluated using Cox regression.
gene expression signature from peripheral blood measured by RNA seq and nano string IO360 | from baseline to surgery and post surgery treatment period, up to 24 months
  The changes of gene expression signature in the peripheral blood from samples collected prior to neoadjuvant treatment and samples collected post-neoadjuvant treatment at each MRI visit will be assessed using paired T-test, and the association between the changes in gene expression signature and clinical outcome (PFS and OS) will be evaluated using Cox regression.
T cell subset and activation markers within peripheral blood measured by flow cytometry | from baseline to surgery and post surgery treatment period, up to 24 months
  The changes of T cell subset and activation markers in the peripheral blood from samples collected prior to neoadjuvant treatment and samples collected post-neoadjuvant treatment at each MRI visit will be assessed using paired T-test, and the association between the changes in T cell subset/activation markers and clinical outcome (PFS and OS) will be evaluated using Cox regression.
TIL quantification including tumor quantification of PD-1, PD-L1, CD3, CD4, CD8, Iba-I, Ki-67 measured by immunohistochemistry of FFPE tissue | from baseline to surgery
  The differences of PD-1, PD-L1, CD3, CD4, CD8, Iba-I, Ki-67 protein expression level between the archival tumor (collected pre-treatment) and protocol tumor (collected post-neoadjuvant treatment) will be assessed using paired T-test, and the association between the changes in the protein expression level and clinical outcome (PFS and OS) will be evaluated using Cox regression.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy F Cloughesy, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- Quan, Los Angeles, California, United States